CLINICAL TRIAL: NCT00716014
Title: A Single-Center, Placebo-Controlled, Rising Dose to Tolerance and Safety Study of TD101, an siRNA Designed for Treatment of Pachyonychia Congenita
Brief Title: Study of TD101, a Small Interfering RNA (siRNA) Designed for Treatment of Pachyonychia Congenita
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pachyonychia Congenita Project (Other)
Responsible Party: Sancy Leachman/Principal Investigator, PC Project
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24013
Record Dates: First submitted 2008-07-15; First posted 2008-07-16 (Estimated); Last update posted 2008-11-19 (Estimated); Status verified 2008-11

CONDITIONS: Pachyonychia Congenita
Keywords: Pachyonychia Congenita; siRNA
MeSH Terms: conditions — Pachyonychia Congenita | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Foot 1 (Active Comparator): An active drug injection of TD101 is injected into a callus on the bottom of one foot.
  Interventions: Drug: TD101
- Foot 2 (Placebo Comparator): An injection of placebo (normal saline) is injected into a callus on the bottom of one foot.
  Interventions: Drug: Normal saline (placebo)

INTERVENTIONS:
Drug: TD101 — TD101 is injection into a callus on the bottom of one of the patient's feet
  Arms: Foot 1
Drug: Normal saline (placebo) — A normal saline solution (placebo) is injected into one of the patient's feet.
  Arms: Foot 2

SUMMARY:
Pachyonychia congenita (PC) is a rare, autosomal dominant keratin disorder affecting the nails, skin, oral mucosae, larynx, hair and teeth. Pathogenic mutations in keratin K6a, K6b, K16 or K17 act via a dominant negative mechanism, leading to manifestations of the disease. The most disabling PC symptom is a painful plantar blistering and keratoderma that requires use of ambulation devices in more than 50 percent of patients. Despite our understanding of the molecular basis of PC, current treatment is limited to mechanical removal of the thick calluses, non-specific topical keratolytics, and oral retinoids, none of which alleviates blistering or plantar pain satisfactorily. A public charity, PC Project, has been founded to support the development of treatments for PC (www.pachyonychia.org). In collaboration with this charity, a small company, TransDerm, Inc., has developed a small interfering RNA (siRNA) that specifically targets a mutation in one of the PC keratins, K6a. As this siRNA targets a single nucleotide mutation, it will only be effective against PC subjects harboring this specific mutation. There are currently only six known patients who carry this mutation in the International Pachyonychia Congenita Research Registry, but three of these patients live in Salt Lake City (a mother and two of her children). We propose to perform a Phase Ib clinical trial to test the safety and tolerability of TD101 in PC patients carrying an N171K mutation. We will complete treatment of the adult patient prior to recruitment of the minors.

ELIGIBILITY:
Inclusion Criteria:

* A positive genetic identification of the N171K mutation in the keratin 6a gene from a CLIA certified laboratory;
* Witnessed, signed informed consent approved by Institutional Review Board/Ethics Committee;
* A signed Health Information Portability and Accountability Act (HIPAA) authorization form which permits the use and disclosure of patient's individually identifiable health information for those enrolled in the United States of America;
* Male or female subjects of any race 10 years of age and older;
* Complete physical examination and medical history indicating no abnormalities that will interfere with study objectives;
* Normal or not clinically significant baseline laboratory tests, including hemogram, ANA, serum chemistry panel, urinalysis, C3a, Bb, and APTT,PT;
* Negative pregnancy test (females only).

Exclusion Criteria:

* Females of childbearing potential not using a highly effective method of birth control (e.g. implants, injectables, combined oral contraceptives, some intrauterine contraceptive devices) during the study;
* Diabetes mellitus requiring treatment other than diet and exercise;
* Treatment of any type for cancer within the last six months;
* History of any significant internal disease;
* Subjects who are known to be allergic to any of the test product(s) or any components in the test product(s) or history of hypersensitivity or allergic reactions to any of the study preparations;
* History of street drug or alcohol abuse;
* Any patient not able to meet the study attendance requirements;
* Subjects who have participated in any other trial of an investigational drug or device within 60 days prior to enrollment or participation in a research study concurrent with this study.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Determine safety/toxicity of TD101 | 18 weeks, followed by 3-month wash out period

SECONDARY OUTCOMES:
Determine efficacy of TD101 | 18 weeks, followed by 3-month wash out period

CONTACTS AND LOCATIONS:
Overall Officials: Sancy A Leachman, MD, PhD, Principal Investigator — PC Project
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States